CLINICAL TRIAL: NCT04152863
Title: A Phase 2, Randomized Clinical Study of Intravenous or Intratumoral Administration of V937 in Combination With Pembrolizumab (MK-3475) Versus Pembrolizumab Alone in Participants With Advanced/Metastatic Melanoma
Brief Title: Efficacy, Safety, and Tolerability of Gebasaxturev (V937) Administered Intravenously or Intratumorally With Pembrolizumab (MK-3475) Versus Pembrolizumab Alone in Participants With Advanced/Metastatic Melanoma (V937-011)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V937-011; V937-011 (Other: Merck Id); 2019-002034-36 (EudraCT Number)
Record Dates: First submitted 2019-11-04; First posted 2019-11-05 (Actual); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Advanced/Metastatic Melanoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2); Coxsackievirus A21; Intracellular Adhesion Molecule-1 (ICAM-1)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IV Gebasaxturev + Pembrolizumab (Experimental): Participants receive gebasaxturev at a dose of 1 X 10^9 TCID50 by IV infusion on Days 1, 3, 5, and 8 of Cycle 1 (28-day cycle) and Day 1 of Cycles 2-8 (21-day cycles) plus pembrolizumab 200 mg by IV infusion on Day 8 of Cycle 1 (28-day cycle) and Day 1 of each subsequent 21-day cycle. Gebasaxturev will be administered for up to 8 cycles (up to 6 months). Pembrolizumab will be administered for up to 35 cycles (up to 2 years).
  Interventions: Biological: Gebasaxturev IV; Drug: Pembrolizumab
- ITu Gebasaxturev + Pembrolizumab (Experimental): Participants receive gebasaxturev at a dose of 3 X 10^8 TCID50 by ITu injection on Days 1, 3, 5, and 8 of Cycle 1 (28-day cycle) and Day 1 of Cycles 2-8 (21-day cycles) plus pembrolizumab 200 mg by IV infusion on Day 8 of Cycle 1 (28-day cycle) and Day 1 of each subsequent 21-day cycle. Gebasaxturev will be administered for up to 8 cycles (up to 6 months). Pembrolizumab will be administered for up to 35 cycles (up to 2 years).
  Interventions: Biological: Gebasaxturev ITu; Drug: Pembrolizumab
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg by IV infusion on Day 8 of Cycle 1 (28-day cycle) and Day 1 of each subsequent 21-day cycle. Pembrolizumab will be administered for up to 35 cycles (up to 2 years).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Biological: Gebasaxturev IV — Administered as an IV infusion of 1 X 10^9 TCID50
  Other Names: Coxsackievirus A21 (CVA21); Formerly known as CAVATAK®; CAV21; V937
  Arms: IV Gebasaxturev + Pembrolizumab
Biological: Gebasaxturev ITu — Administered as an ITu injection of 3 X 10^8 TCID50
  Other Names: Coxsackievirus A21 (CVA21); Formerly known as CAVATAK®; CAV21; V937
  Arms: ITu Gebasaxturev + Pembrolizumab
Drug: Pembrolizumab — Administered as an IV infusion of 200 mg
  Other Names: MK-3475; Keytruda®

SUMMARY:
This is a Phase 2 study to assess the efficacy, safety, and tolerability of gebasaxturev administered both intratumorally (ITu) and intravenously (IV) as combination therapy with pembrolizumab (MK-3475) versus pembrolizumab alone in anti-programmed cell death ligand 1 (anti-PD-L1)-treatment-naive participants with advanced/metastatic melanoma. The primary hypothesis of the study is that gebasaxturev administered either ITu or IV in combination with pembrolizumab results in a superior objective response rate (ORR) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) based on blinded independent central review (BICR), compared to pembrolizumab alone. This study will be terminated once all participants finish treatment with V937. Participants eligible to continue to receive pembrolizumab will be transferred to MK-3475-587 study.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed diagnosis of advanced/metastatic melanoma.
* Has Stage III or Stage IV melanoma.
* Must be naive to anti-PD-L1 treatment, talimogene laherparepvec (TVEC) and other oncolytic viruses.
* Has 2 lesions as defined below:

  * At least 1 cutaneous or subcutaneous lesion that is amenable to IT injection and biopsy and measurable per RECIST 1.1
  * At least 1 distant and/or discrete noninjected lesion that is amenable to biopsy and measurable per RECIST 1.1
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Demonstrates adequate organ function
* Male participants refrain from donating sperm during the intervention period and for at least 120 days after the last dose of study intervention PLUS are either abstinent from heterosexual intercourse OR agree to use approved contraception during that period
* Female participants are not pregnant or breastfeeding and are not a woman of childbearing potential (WOCBP) OR are a WOCBP that agrees to use contraception during the treatment and for at least 120 days after the last dose of study intervention
* Has measurable disease per RECIST 1.1
* Is able to provide newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Human Immunodeficiency Virus (HIV)-infected participants must have well controlled HIV on anti-retroviral therapy (ART), defined as:

  * Must have Cluster of Differentiation 4 (CD4)+ T-cell count >350 cells/mm^3 at time of screening
  * Must have achieved and maintained virologic suppression
  * Must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to study entry
  * The combination ART regimen must not contain any antiretroviral medication other than abacavir, dolutegravir, emtricitabine, lamivudine, raltegravir, rilpivirine, or tenofovir

Exclusion Criteria:

* Has had chemotherapy, definitive radiation, or biological cancer therapy or an investigational agent or investigational device within 4 weeks prior to the first dose of study intervention or has not recovered to Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 or better from any AEs that were due to cancer therapeutics administered more than 4 weeks earlier
* Has ocular melanoma
* Has radiographic evidence of major blood vessel infiltration
* Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug
* Has an active autoimmune disease that has required systemic treatment in the past 2 years except vitiligo or resolved childhood asthma/atopy
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the study requirements
* Has undergone allogeneic hematopoietic stem cell transplantation within the last 5 years
* Has not fully recovered from major surgery without significant detectable infection
* Active cardiovascular disease (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure or serious cardiac arrhythmia requiring medication
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or other agents such as cytotoxic T-lymphocyte-associated protein-4 (CTLA-4), OX-40, Cluster of Differentiation 137 (CD137)
* Has received a live vaccine within 30 days prior to the first dose of study drug
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy in excess of replacement doses or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has hypersensitivity to pembrolizumab and/or any of its excipients
* Has hypersensitivity to gebasaxturev or any of its excipients
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of Hepatitis B or known active Hepatitis C virus infection
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (30):
- United States (4):
  - Henry Ford Hospital ( Site 0008), Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey ( Site 0002), New Brunswick, New Jersey
  - Providence Portland Medical Center [Portland, OR] ( Site 0005), Portland, Oregon
  - Northwest Medical Specialties, PLLC ( Site 0006), Tacoma, Washington
- Australia (3):
  - The Queen Elizabeth Hospital ( Site 0143), Woodville, South Australia
  - Alfred Health ( Site 0142), Melbourne, Victoria
  - Fiona Stanley Hospital ( Site 0141), Murdoch, Western Australia
- Chile (2):
  - FALP-UIDO ( Site 2062), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 2061), Santiago, Region M. de Santiago
- France (2):
  - Centre Georges Francois Leclerc ( Site 2025), Dijon, Cote-d Or
  - CHU de Grenoble Hopital Nord ( Site 2027), La Tronche, Isere
- Germany (3):
  - Universitaetsklinikum Tuebingen-Hautklinik ( Site 2001), Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Regensburg ( Site 2007), Regensburg, Bavaria
  - Universitaetsklinikum Leipzig AOeR ( Site 2005), Leipzig, Saxony
- Israel (3):
  - Rambam Health Care Campus-Oncology Division ( Site 0040), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0042), Jerusalem
  - Chaim Sheba Medical Center ( Site 0041), Ramat Gan
- Italy (2):
  - Istituto Europeo di Oncologia ( Site 2040), Milan
  - Policlinico Le Scotte - A.O. Senese ( Site 2039), Siena
- Oslo Universitetssykehus Radiumhospitalet ( Site 0060), Oslo, Norway
- South Africa (5):
  - WITS Clinical Research CMJAH Clinical Trial Site ( Site 0101), Johannesburg, Gauteng
  - Clinical Research Unit - University of Pretoria ( Site 0102), Pretoria, Gauteng
  - Wilgers Oncology Centre ( Site 0103), Pretoria, Gauteng
  - Little Company of Mary Hospital ( Site 0100), Pretoria, Gauteng
  - Cape Town Oncology Trials Pty Ltd ( Site 0104), Cape Town, Western Cape
- South Korea (2):
  - Seoul National University Hospital ( Site 1992), Seoul
  - Severance Hospital Yonsei University Health System ( Site 1993), Seoul
- Spain (3):
  - Onkologikoa - Instituto Oncologico de San Sebastian ( Site 0088), Donostia / San Sebastian, Gipuzkoa
  - Clinica Universitaria de Navarra. ( Site 0082), Pamplona, Navarre
  - Hospital Clinico Universitario de Valencia ( Site 0090), Valencia, Valenciana, Comunitat

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Deng JZ, Rustandi RR, Barbacci D, Swartz AR, Gulasarian A, Loughney JW. Reverse-Phase Ultra-Performance Chromatography Method for Oncolytic Coxsackievirus Viral Protein Separation and Empty to Full Capsid Quantification. Hum Gene Ther. 2022 Jul;33(13-14):765-775. doi: 10.1089/hum.2022.013. Epub 2022 Jun 1. PMID 35387488
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Intravenous (IV) Gebasaxturev + IV Pembrolizumab: Participants received gebasaxturev at a dose of 1 X 10^9 50% tissue culture infectious dose (TCID50) by IV infusion on Days 1, 3, 5, and 8 of Cycle 1 (28-day cycle) and Day 1 of Cycles 2-8 (21-day cycles) plus pembrolizumab 200 mg by IV infusion on Day 8 of Cycle 1 (28-day cycle) and Day 1 of each subsequent 21-day cycle. Gebasaxturev was administered for up to 8 cycles (up to 6 months). Pembrolizumab was administered for up to 35 cycles (up to 2 years).
- Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab: Participants received gebasaxturev at a dose of 3 X 10^8 TCID50 by ITu injection on Days 1, 3, 5, and 8 of Cycle 1 (28-day cycle) and Day 1 of Cycles 2-8 (21-day cycles) plus pembrolizumab 200 mg by IV infusion on Day 8 of Cycle 1 (28-day cycle) and Day 1 of each subsequent 21-day cycle. Gebasaxturev was administered for up to 8 cycles (up to 6 months). Pembrolizumab was administered for up to 35 cycles (up to 2 years).
- Pembrolizumab IV: Participants received pembrolizumab 200 mg by IV infusion on Day 8 of Cycle 1 (28-day cycle) and Day 1 of each subsequent 21-day cycle. Pembrolizumab was administered for up to 35 cycles (up to 2 years).
Period: Overall Study
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Started | 28 | 28 | 29
Treated | 28 | 28 | 26
Completed | 0 | 0 | 0
Not Completed | 28 | 28 | 29
Not completed — Death | 13 | 12 | 7
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Participation in Study Terminated by Sponsor | 12 | 14 | 18
Not completed — Withdrawal by Subject | 2 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV | Total
Number analyzed (Participants) | 28 | 28 | 29 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (10.5) | 58.3 (13.6) | 60.5 (11.9) | 61.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 11 | 29
  Male | 20 | 18 | 18 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 3 | 11
  Not Hispanic or Latino | 25 | 21 | 26 | 72
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 3 | 2 | 8
  White | 23 | 24 | 26 | 73
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Cancer M Staging at Baseline [Count of Participants; unit: Participants] — Randomization was stratified based on 4 metastatic melanoma subsets: M1a (nonvisceral (distant cutaneous, subcutaneous, nodal); M1b (lung); M1c (noncentral nervous system (CNS) visceral); and M1d (involves the CNS), as defined by the AJCC (American Joint Committee on Cancer) Cancer Staging Manual, Eighth Edition. M1c and M1d have different prognoses compared to M1a and M1b, warranting stratification.
  Participants
    M1a | 7 | 9 | 9 | 25
    M1b | 6 | 3 | 5 | 14
    M1c | 12 | 14 | 9 | 35
    M1d | 1 | 1 | 1 | 3
    Missing | 2 | 1 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants who experienced a Complete Response (CR: disappearance of all lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions, without evidence of progression based on non-target or new lesions) as assessed by BICR per RECIST 1.1 which was modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a CR or PR based on modified RECIST 1.1 is presented.
Time Frame: Up to ~ 35 months
Population: All allocated participants included in the treatment group to which they were allocated.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 28 | 28 | 29
Percentage of Participants | 46.4 [30.1 to 63.4] | 39.3 [23.8 to 56.5] | 34.5 [20.0 to 51.4]
Statistical Analysis 1: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Superiority; p = 0.1812, Stratified Miettinen & Nurminen method; To ensure adequate number of participants, strata were combined according to sSAP when one treatment had 0 participants in a particular stratum; Mean Difference (Net) = 11.9, 90% CI 2-sided [-9.5 to 32.5]
Statistical Analysis 2: Comparison: Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Superiority; p = 0.3548, Stratified Miettinen & Nurminen method; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 4.8, 90% CI 2-sided [-16.2 to 25.5]
Statistical Analysis 3: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in % = 7.1, 90% CI 2-sided [-14.6 to 28.2]

2. Secondary Outcome: Progression Free Survival (PFS) Per RECIST 1.1 as Assessed by BICR
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD.
Time Frame: Up to ~ 35 months
Population: All allocated participants included in the treatment group to which they were allocated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 28 | 28 | 29
Months | 12.7 [2.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 7.3 [2.7 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 8.6 [2.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.50 to 2.27]
Statistical Analysis 2: Comparison: Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.51 to 2.29]
Statistical Analysis 3: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.50 to 2.04]

3. Secondary Outcome: Duration of Response (DOR)
Description: For participants who demonstrated a confirmed complete response (CR: disappearance of all lesions) or confirmed Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions, without evidence of progression based on non-target or new lesions.) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurred first. RECIST 1.1 was adjusted for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ and was assessed by BICR for this outcome measure.
Time Frame: Up to ~ 35 months
Population: All allocated participants included in the treatment group to which they were allocated.
Measure: Median (Full Range); unit: Months
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 13 | 11 | 10
Months | NA [NA to NA] — NA = Median, upper and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [4.1 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper and lower limit not reached at time of data cut-off due to insufficient number of participants with an event.

4. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1, as Assessed by the Investigator
Description: ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 as assessed by the investigator modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a CR or PR based on modified RECIST 1.1 was presented.
Time Frame: Up to ~ 35 months
Population: All allocated participants included in the treatment group to which they were allocated.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 28 | 28 | 29
Percentage of Participants | 39.3 [23.8 to 56.5] | 39.3 [23.8 to 56.5] | 41.4 [25.9 to 58.3]
Statistical Analysis 1: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in percentage = -2.1, 90% CI 2-sided [-23.1 to 19.2]
Statistical Analysis 2: Comparison: Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in percentage = -2.1, 90% CI 2-sided [-23.1 to 19.2]
Statistical Analysis 3: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab; Test type: Other — Difference in percentage based on Miettinen & Nurminen method; Difference in % = 0.0, 90% CI 2-sided [-21.2 to 21.2]

5. Secondary Outcome: Progression Free Survival (PFS) RECIST 1.1, as Assessed by the Investigator
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1 as assessed by the investigator, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD.
Time Frame: Up to ~ 35 months
Population: All allocated participants included in the treatment group to which they were allocated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 28 | 28 | 29
Months | 4.6 [2.4 to 15.3] | 6.5 [2.7 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 15.4 [2.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.70 to 3.02]
Statistical Analysis 2: Comparison: Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [0.62 to 2.68]
Statistical Analysis 3: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.60 to 2.22]

6. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1, as Assessed by the Investigator
Description: For participants who demonstrated a confirmed complete response (CR: disappearance of all lesions) or confirmed Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by the investigator, DOR was defined as the time from first documented evidence of CR or PR until disease progression or death.
Time Frame: Up to ~ 35 months
Population: All allocated participants included in the treatment group to which they were allocated.
Measure: Median (Full Range); unit: Months
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 11 | 11 | 12
Months | NA [7.1 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [NA to NA] — NA = Median, upper and lower limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [8.4 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.

7. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from randomization to death due to any cause.
Time Frame: Up to ~ 35 months
Population: All allocated participants included in the treatment group to which they were allocated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 28 | 28 | 29
Months | 17.5 [6.8 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | 24.1 [11.4 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of participants with an event. | NA [14.0 to NA] — NA = Median and upper limit not reached at time of data cut-off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.71 to 3.79]
Statistical Analysis 2: Comparison: Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab vs Pembrolizumab IV; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.47 to 2.68]
Statistical Analysis 3: Comparison: Intravenous (IV) Gebasaxturev + IV Pembrolizumab vs Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab; Test type: Other — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [0.64 to 3.02]

8. Secondary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to ~ 37 months
Population: All randomized participants who received at least one dose of study medication. Participants were analyzed in the treatment arm corresponding to the study treatment they actually received.
Measure: Number; unit: Percentage of Participants
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 28 | 28 | 26
Percentage of Participants | 100 | 100 | 84.6

9. Secondary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 8
Time Frame: Up to ~ 27 months
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
Number analyzed (Participants) | 28 | 28 | 26
Percentage of Participants | 14.3 | 7.1 | 3.8

ADVERSE EVENTS:
Time Frame: Up to ~ 37 months
Description: All-cause mortality (ACM) was analyzed in all randomized participants. Safety analyses were conducted in all randomized participants who received at least 1 dose of study intervention. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study treatment. Thus, MedDRA 26.0 preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded.
Arm/Group | Intravenous (IV) Gebasaxturev + IV Pembrolizumab | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab | Pembrolizumab IV
All-Cause Mortality (participants affected / at risk) | 14/28 | 12/28 | 9/29
Serious Adverse Events (participants affected / at risk) | 8/28 | 5/28 | 4/26
Other Adverse Events (participants affected / at risk) | 27/28 | 27/28 | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous (IV) Gebasaxturev + IV Pembrolizumab (N=28) | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab (N=28) | Pembrolizumab IV (N=26)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Overlap syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous (IV) Gebasaxturev + IV Pembrolizumab (N=28) | Intratumoral (ITu) Gebasaxturev + IV Pembrolizumab (N=28) | Pembrolizumab IV (N=26)
Anaemia (Blood and lymphatic system disorders) | 12 (15) | 5 (9) | 7 (8)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 3 (7) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (3) | 1 (3)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 1 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (3) | 1 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 0 (0) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (6) | 3 (3) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (4)
Constipation (Gastrointestinal disorders) | 6 (8) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 3 (4)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (10) | 5 (6) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (6) | 0 (0) | 2 (2)
Asthenia (General disorders) | 2 (3) | 3 (4) | 3 (3)
Axillary pain (General disorders) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 8 (8) | 11 (11) | 6 (7)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 0 (0)
Xerosis (General disorders) | 1 (1) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 3 (5) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (4)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (5) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (8) | 5 (11) | 9 (14)
Aspartate aminotransferase increased (Investigations) | 5 (8) | 3 (5) | 4 (6)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 3 (6) | 4 (5)
Blood bilirubin increased (Investigations) | 1 (4) | 1 (2) | 2 (4)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Blood creatinine increased (Investigations) | 3 (7) | 1 (1) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 4 (6) | 2 (2) | 4 (4)
Blood thyroid stimulating hormone increased (Investigations) | 2 (3) | 3 (3) | 3 (5)
Weight decreased (Investigations) | 7 (7) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 3 (3) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (5) | 2 (2) | 1 (5)
Hyperphosphataemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (8) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (5) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 5 (6) | 1 (1) | 4 (5)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 6 (9) | 5 (8)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 5 (5) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 3 (3)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 5 (7) | 5 (6)

LIMITATIONS AND CAVEATS:
This study was terminated due to the sponsor's development decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT04152863/Prot_SAP_001.pdf